CLINICAL TRIAL: NCT02278237
Title: Pre/Post Pilot Test of VME for the Video vs. TTG Respiratory Inhaler Technique Assessment and InstructioN Study
Brief Title: Pre/Post Pilot Test of Video Module Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB12-1844
Record Dates: First submitted 2014-10-10; First posted 2014-10-29 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VME Group (Experimental): Pre and post VME education group. The Intervention is the use of the virtual education module rather than the interpersonal educational strategy.
  Interventions: Behavioral: VME Group

INTERVENTIONS:
Behavioral: VME Group — Received inhaler education through VME (virtual education module)
  Other Names: Video Module Education (VME)

SUMMARY:
Asthma and Chronic obstructive pulmonary disease (COPD) results in over a million hospitalizations in the United States annually and COPD is the third leading cause of 30-day re-hospitalizations. Clinical trials have established the efficacy of treatments primarily dispensed via respiratory inhaler devices that reduce morbidity and health care utilization if they are used correctly. The effectiveness of these medications in real-world settings is limited by the fact that patients often do not use inhalers correctly. Current guidelines recommend assessing and teaching inhaler technique at all health care encounters, including hospitalization. Over 75% of hospitalized patients in an urban, predominantly underserved population misused their respiratory inhalers, highlighting a missed opportunity to educate these patients with high potential to benefit. Hospitalization, therefore, provides a potential 'teachable moment' to correct this misuse. My preliminary data indicate that one strategy, in-person teach-to-goal (TTG), is effective in teaching hospitalized patients proper inhaler technique and is more effective than simple verbal instruction. While TTG is a promising, several limitations prevent widespread adoption. TTG is time-consuming and costly. Also, reinforcement may be needed, which may be impractical with in-person TTG. One potential method to surmount TTG's limitations is use of interactive video module education (VME) that has the potential to be less costly, maintain fidelity, and be more easily extended into the post-discharge setting than in-person TTG. Before widespread implementation of VME, it is critical to rigorously develop and test VME for inhaler education in the hospital setting. Ultimately, it will also be important to understand patients' ability and willingness to use post-discharge VME for educational reinforcement to allow for this strategy to transition patients across care settings from hospital to home.

We hypothesize that interactive VME will lead to non-inferior rates of ability to demonstrate correct inhaler use compared to rates with TTG among hospitalized patients with Asthma or COPD.

For this study we are testing the preliminary efficacy of VME to teach respiratory inhaler technique prior to implementing a larger RCT to test the comparative effectiveness of VME versus TTG.

DETAILED DESCRIPTION:
The specific aim to test this hypothesis is:

To iteratively test VME to teach correct use of metered dose inhaler (MDIs) and dry-powder Diskus® devices to hospitalized patients with Asthma or COPD. We partnered with software development companies to develop VME modules that (self)-assess and teach respiratory inhaler technique to hospitalized participants. We have tested the VME in focus groups. Now that the VME is developed we will iteratively pilot test (n=30-40) the VME strategy (up to 3 rounds (90-120 total)) to obtain important patient feedback,preferences and preliminary efficacy estimates for the module.

We hypothesize that participants' post-VME inhaler technique will be significantly better than their pre-VME inhaler technique.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older
2. Admission to the inpatient medical service and surgical service
3. Physician-diagnosed COPD or asthma. We will enroll patients even if the primary reason for admission is not COPD or asthma (e.g., patients admitted for heart failure, but with a physician diagnosis of COPD are eligible).

Exclusion Criteria:

1. Currently in an intensive care unit
2. Physician declines to provide consent
3. Patient unable to provide consent (e.g., history of cognitive impairment, unable to understand English) or declines to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie G. Press, MD, MPH, Principal Investigator — University of Chicago

RESULTS

PARTICIPANT FLOW:
Groups:
- VME Group: Video Module Education (VME): The RE will provide participants with a tablet device and will demonstrate how to access VME and complete the pre/post e-learning assessments. The RE will provide technical support but will neither participate directly in the education nor help with the self-assessments. The participants will first complete the pre-assessment e-learning tool on the tablet. They will then watch the video instruction that will provide a complete demonstration with verbal instructions on correct inhaler technique. Next the participants will complete the post-assessment e-learning tool. Based on participants' performance, they will be directed to further tailored video-instruction. The cycle of self-assessment and video instruction will continue until sufficient mastery has been achieved.
Period: Overall Study
Arm/Group | VME Group
Started | 90
Completed | 83
Not Completed | 7

BASELINE CHARACTERISTICS:
Groups:
- VME Group: Video Module Education (VME)
Arm/Group | VME Group
Number analyzed (Participants) | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 79
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Inhaler Misuse Pre- and Post-VME
Description: Assess patient's inhaler technique using Inhaler checklists by the trained assessor.
  The primary outcome will be comparing post-intervention to pre-intervention scores; secondary outcome will be 30 days post-discharge visit
  We will define inhaler technique in two ways:
  1. Correct Use (i.e., >75% of steps correct)
  2. Mastery (i.e., perfect technique, 100% steps correct)
Time Frame: Up to 30 days
Measure: Number; unit: participants
Arm/Group | VME Group
Number analyzed (Participants) | 83
participants
  Misuse pre-VME | 83
  Misuse post-VME | 24

2. Secondary Outcome: Symptom Burden
Description: Assess patient's respiratory symptoms/morbidity, which includes the Borg symptom score, Asthma Symptom Severity Index (ASSI), Chronic Bronchitis Symptom Questionnaire, COPD Severity Score (CSS), Airway Questionnaire (AQ-20), COPD Helplessness Index (CHI) and demographic and other clinical information.
Time Frame: up to 30 days
Reporting Status: Not Posted

3. Secondary Outcome: Quality of Life (QOL)
Description: Use validated disease specific QOL tools (i.e., asthma or COPD QOL tools)
Time Frame: up to 30 days
Reporting Status: Not Posted

4. Secondary Outcome: Self-efficacy of Inhaler Technique
Description: Assess patient's confidence in using their inhalers.
  We will ask patients to report if they: strongly disagree/disagree/neutral/agree/strongly agree with the statement: "I am confident that I know how to use this respiratory inhaler correctly".
Time Frame: up to 30 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through study completion, which was up to 30 days.
Description: Based on the nature of the study, we foresee that the risk for participation does not exceed the risks of typical daily activities. We expect that a patient's All-Cause Mortality does not change based on their inclusion in this study.
Arm/Group | VME Group
All-Cause Mortality (participants affected / at risk) | 0/90
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes